CLINICAL TRIAL: NCT00003362
Title: Pilot Trial of Multi-Epitope Melanoma Peptide Vaccine Using GM-CSF, Montanide and QS-21 as Adjuvants
Brief Title: Vaccine Therapy Plus Immune Adjuvants in Treating Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 98-012; CDR0000066345 (Registry Identifier: PDQ (Physician Data Query)); NCI-T97-0110
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — saponin QA-21V1; incomplete Freund's adjuvant; sargramostim

INTERVENTIONS:
Biological: QS21
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from peptides that are found on melanoma cells may make the body build an immune response and kill melanoma cells. Combining vaccine therapy with immune adjuvants, such as GM-CSF, Montanide ISA-51, or QS21, may be a more effective treatment for advanced melanoma.

PURPOSE: Randomized phase II trial to study the effectiveness of gp 100-tyrosinase peptide vaccine with one of the immune adjuvants GM-CSF, Montanide ISA-51, or QS21 in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the immunogenicity of gp100-tyrosinase peptide vaccine with sargramostim (GM-CSF), Montanide ISA-51, or QS21 as adjuvant in patients with advanced melanoma. II. Determine the toxicity of this multiepitope melanoma peptide vaccine in conjunction with these 3 adjuvants in these patients. III. Evaluate the antitumor effects of this multiepitope melanoma peptide vaccine in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to age (65 years and under vs more than 65 years) and previous systemic chemotherapy (yes vs no). Patients are randomized to 1 of 3 treatment arms: Arm I (Sargramostim (GM-CSF) as adjuvant): Patients receive 3 monthly vaccinations with gp100-tyrosinase peptide vaccine administered intradermally during weeks 1, 5, and 9. For each vaccination, GM-CSF is administered intradermally on days 1-10; the vaccine is administered on day 7. Arm II (Montanide ISA-51): Patients receive 3 monthly vaccinations with gp100-tyrosinase peptide vaccine mixed with Montanide ISA-51 and administered subcutaneously (SQ) during weeks 1, 5, and 9. Arm III (QS21 as adjuvant): Patients receive 3 monthly vaccinations with gp100-tyrosinase peptide vaccine mixed with QS21 and administered SQ during weeks 1, 5, and 9. Patients with stable or responding disease may receive 3 additional monthly immunizations beginning 3-6 months following completion of 1 course of immunizations if there is evidence of T cell response against either wild type peptide. Patients are followed at weeks 13 and 17.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable stage III or stage IV melanoma Patients who are disease free following surgical resection or chemotherapy for stage III or IV disease also eligible HLA-A201 positive

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 5 months Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 75,000/mm3 LDH no greater than 2 times upper limit of normal No active bleeding Hepatic: Albumin at least 3.5 mg/dL Renal: Not specified Other: Not pregnant or less than 3 months postpartum Fertile patients must use effective contraception No serious underlying medical conditions No known immunodeficiency No active infection No retinal or choroidal eye disease

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered No prior tyrosinase or gp100 peptides No prior Montanide ISA-51 No prior melanoma protein vaccine or melanoma whole cell vaccines No other concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No concurrent chemotherapy Endocrine therapy: At least 2 weeks since prior systemic steroids and recovered No concurrent systemic steroids Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to the spleen No concurrent radiotherapy Surgery: Recovered from any prior surgery No prior splenectomy Other: At least 1 week since prior antiinflammatory drugs and recovered At least 1 week since prior antihistamines and recovered No concurrent antiinflammatory drugs No concurrent antihistamines No concurrent antimicrobial drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Chapman, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States